CLINICAL TRIAL: NCT03943108
Title: Criticality Analysis of Diabetic Gait Within the PAIDOS Pediatric Clinic for Obese Children (PAIDOS: Pediatric Attention Integral and Dynamic for Obese Children Program)- A Feasibility Study
Brief Title: Criticality Analysis of Diabetic Gait Within a Primary Care Pediatric Clinic for Obese Children (PAIDOS)
Acronym: PAIDOS
Status: Completed | Type: Observational
Sponsor: Dr Salvador Villalpando-Carrion (Other)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Sponsor-Investigator, Dr Salvador Villalpando-Carrion, Head of Pediatric Gastroenterology and Nutrition, Hospital Infantil de Mexico Federico Gomez
Organization: Hospital Infantil de Mexico Federico Gomez (Other)
Other Study IDs: HIM-060-09
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2019-09

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese teenagers within the PAIDOS clinic: Obese children within the PAIDOS clinic, Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico.
  Interventions: Diagnostic Test: Gait analysis
- Healthy children: Healthy children living in Mexico City, Mexico.
  Interventions: Diagnostic Test: Gait analysis
- Children with Type 2 Diabetes: Chjildren with Type 2 Diabetes attending the Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico.
  Interventions: Diagnostic Test: Gait analysis

INTERVENTIONS:
Diagnostic Test: Gait analysis — Gait recorded using a sensor on the 4th vertebrae of the lumbar spine, once a week across 6 weeks during the routine PAIDOS clinic. Critical changes in walking control, stride frequency and length will be observed as individuals change speed; effectively stressing their mobility.

SUMMARY:
One of the difficulties with diabetes care is the problem of predicting progression to more severe stages using current measures (for example blood glucose, HbA1c). This feasibility study aims to use Criticality Analysis (CA) of gait to monitor the progression of the condition as well as identifying individuals at risk of developing diabetes among children in Mexico.The study will investigate whether gait analysis can be used as a fast, reliable and cost effective way to detect individuals at risk of developing Type 2 Diabetes (T2DM) as early treatment could reduce the number of cases that develop into full T2DM.

DETAILED DESCRIPTION:
This feasibility study aims to the do the following:

1. To evaluate the use of Criticality Analysis of Gait as means of Diabetes assessment.
2. To design and set up a clinical feasibility study in a hospital (Hospital Infantil de Mexico) with adolescent patients on different clinical stages of type 2 Diabetes mellitus (DM).
3. To analyse the collected data and validate Gait data analysis as mechanism for identifying and monitoring pre-diabetic teenagers.
4. To use the feasibility study conducted in Mexico to develop a robust method using Gait analysis for diabetes prevention and management.

Participants will be selected from the Primary Care Pediatric Clinic for Obese Children (PAIDOS) in the Hospital Infantil de México Federico Gómez, Mexico City, Mexico. Sixty participants will be selected and divided into three groups: 40 obese non-diabetic subjects, 10 with Type 2 Diabetes and 10 healthy subjects as controls. Obese participants within the Paidos clinic will undergo standard clinical care that includes dietary prescription of caloric intake according to height, 150 min weekly physical activity, group cognitive-behavioural intervention, 6 session of obesity awareness and educational program.

Gait will be recorded in all groups using a sensor on the 4th vertebrae of the lumbar spine, once a week across 6 weeks during the routine PAIDOS clinic. Critical changes in walking control, stride frequency and length will be observed as individuals change speed; effectively stressing their mobility. The study will be repeated after 3-6 months as a follow up.

Data analysis will be performed in a semi-blind manner in order to test the efficacy of the criticality analysis Rate control of Chaos (RCC) model. In order to provide an objective measure of analysis, the anonymised data will be presented to the nonlinear RCC models, where results can be extracted and compared afterwards to known states.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 95 th percentile for age
* Living in Major Mexico City area

Exclusion Criteria:

* Diabetic patients
* major physical disability

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Individuals attending the Primary Care Pediatric Clinic for Obese Children (PAIDOS) in the Hospital Infantil de Mexico Federico Gomez, living in the Major city area of Mexico City, Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Gait | 6 weeks, 3 and 6 month post-baseline follow-up
  Critical changes in walking control, stride frequency and length observed as individuals change speed using a movement sensor (Inertial Measurement Units (IMU) on the 4th vertebrae of the lumbar spine). Recorded during a 10 metre walk and 6 minute walk test

SECONDARY OUTCOMES:
6 Minute Walk test (6MWT) | 6 weeks, 3 and 6 month post-baseline follow-up
  Distance traveled during the 6MWT in metres
Borg scale of perceived exertion | 6 weeks, 3 and 6 month post-baseline follow-up
  Recorded during the 6MWT
Heart rate | 6 weeks, 3 and 6 month post-baseline follow-up
  Number of beats per minute (BPM) recorded before and after the 6MWT. Determination by palpation of radial, brachial, carotid, or other pulse or by auscultation in precordial area using a stethoscope.
Respiratory rate | 6 weeks, 3 and 6 month post-baseline follow-up
  Recorded before and after the 6MWT.
O2 saturation (mmHg) using a pulse Oximeter | 6 weeks, 3 and 6 month post-baseline follow-up
  Recorded before and after the 6MWT.
Blood Pressure (mmHg) using a baumanometer | 6 weeks, 3 and 6 month post-baseline follow-up
  Recorded before and after the 6MWT
Insulin | 6 weeks, 3 and 6 month post-baseline follow-up
  Measured in microUnit/milliliter (McU/mL) of blood.
Fasting blood Glucose | 6 weeks, 3 and 6 month post-baseline follow-up
  Level of glucose after 12 hours fasting (overnight) measured in milligram/deciliter (mg/dL) of blood.
Hemoglobin A1C | 6 weeks, 3 and 6 month post-baseline follow-up
  Also known as glycated hemoglobin test, and glycohemoglobin. Measured in milligram/deciliter (mg/dL) of blood.
Total cholesterol | 6 weeks, 3 and 6 month post-baseline follow-up
  Measured in milligram/deciliter (mg/dL) of blood.
Level of High-density lipoprotein (HDL) in blood | 6 weeks, 3 and 6 month post-baseline follow-up
  Measured in milligram/deciliter (mg/dL) of blood.
Low-density lipoprotein (LDL) | 6 weeks, 3 and 6 month post-baseline follow-up
  Measured in milligram/deciliter (mg/dL) of blood.
Triglycerides | 6 weeks, 3 and 6 month post-baseline follow-up
  Measured in milligram/deciliter (mg/dL) of blood.
Alanine aminotransferase (ALT) | 6 weeks, 3 and 6 month post-baseline follow-up
  Measured in microUnit/milliliter (McU/mL) of blood.
Aspartate aminotransferase (AST) | 6 weeks, 3 and 6 month post-baseline follow-up
  Measured in millimoles Per Litre (mmol/L).
Homeostatic model assessment (HOMA) Index | 6 weeks, 3 and 6 month post-baseline follow-up
  Index that allows the re-estimation of insulin resistance and Beta cell function through glucose concentration and plasma insulin during fasting state.
Body Mass Index (BMI)- Kg/m2 | 6 weeks, 3 and 6 month post-baseline follow-up
Hip Circumference | 6 weeks, 3 and 6 month post-baseline follow-up
  Maximum perimeter of the hips at the gluteal level in centimeters (cm) using a tape measure.
Waist Circumference | 6 weeks, 3 and 6 month post-baseline follow-up
  Maximum circumference of the horizontal line between the last rib and the superior iliac crest in centimetres (cm) using a tape measure.
Height | Baseline- Week 1
  Centimeters (cm)
Weight | 6 weeks, 3 and 6 month post-baseline follow-up
  Kilograms (Kg)
Leg Length | Baseline- Week 1
  The distance from the anterior superior iliac spine to the medial malleolus in centimetres (cm) using a tape measure.
Shoe Size | Baseline- Week 1
  Mexican Shoe Size (length of foot in centimeters (cm) using a tape measure).
Physical Activity- Accelerometer | 6 weeks
  Axivity AX3 Monitors
Health Behaviour in School Aged Children (HSBC)- Eating Habits Questionnaire | 6 weeks
  Two multiple choice questions. 1 question assesses the frequency of breakfast consumption during weekdays and weekends. For weekdays- scores range from 1 ("I never have breakfast during weekdays") - 6 ("Five days"). For weekends scores range from 1 ("I never have breakfast during the weekend") to 3 ("I usually have breakfast on both weekend days (Saturday AND Sunday)". The higher the score the better the outcome.
  1 question assesses food consumption frequency of fruit, vegetables, sweets and soft drinks that contain sugar.Scores range from 1 ("Never") to 7 ("Every day, more than once"). Higher scores on fruit and vegetables = better outcome. The higher the score on sweets and soft drinks the worse the outcome.

OTHER OUTCOMES:
Single item enjoyment of physical activity scale | 6 weeks, 3 and 6 month post-baseline follow-up
  During each clinic visit the participant will be asked the following, single answer question (translated into Spanish):
  How much would you agree with the following? "I enjoy being physically active"
  The answer is a seven point scale ranging from 1 (Strongly Disagree) to 7 (Strongly Agree). The higher the score the better the outcome.
Fatigue | 6 weeks, 3 months, 6 months
  The children will be asked the following question to assess fatigue levels (translated into spanish):
  "On average, what fraction of the day do you feel tired or very tired?"
  1) None/nothing, 2) A quarter of the day, 3) Half of the day, 4) Three quarters of the day, 5) All of the day
  The higher the score the worse the fatigue outcome.
Self-reported Physical activity- completion of daily exercise | 6 weeks, 3 months, 6 months
  The children are asked whether they have completed their daily exercise using an online survey (as part of the PAIDOS program). The following is translated into Spanish:
  Have you completed the activity / exercises today? Yes/No
Self-reported Physical activity- reason for no completion | 6 weeks, 3 months, 6 months
  The children are asked the reason for not completing their daily exercise using an online survey (as part of the PAIDOS program). The following question is translated into Spanish:
  If you have answered no, indicate why:
  1. I was sick
  2. My muscles or joints hurt
  3. Today was one of my days of rest
  4. I had an event
  5. I did not want to do it (indicate the reason)
Self-reported Physical activity- type of daily exercise | 6 weeks, 3 months, 6 months
  The children are asked the type of exercise they did that day using an online survey (as part of the PAIDOS program). The following open text box question is translated into Spanish:
  What physical activity did you do today?
Self-reported Physical activity- time spent doing daily exercise | 6 weeks, 3 months, 6 months
  The children are asked the time spent doing the exercise in minutes using an online survey (as part of the PAIDOS program). The following question is translated into Spanish:
  How much time did you spend doing this physical activity in minutes?
  Higher number of minutes equals a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Arantza Aldea, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Hospital Infantil de Mexico, Mexico City, Mexico